CLINICAL TRIAL: NCT01922024
Title: Detection of Microorganisms and Antibiotic Resistance Genes in Lower Respiratory Tract (LRT) Samples Using the Curetis Unyvero LRT55 Application
Brief Title: Detection of Microorganisms and Antibiotic Resistance Genes Using the Curetis Unyvero LRT55 Application
Acronym: LRT55
Status: Completed | Type: Observational
Sponsor: Curetis GmbH (Industry)
Collaborators: Global BioClinical (Industry)
Responsible Party: Sponsor
Other Study IDs: CURETIS LRT55 Study - V 6.0
Record Dates: First submitted 2013-08-07; First posted 2013-08-14 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchial lavage (BAL) Tracheal aspirate (TA)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prospective Fresh Clinical Specimens: Patients with suspicion of lower respiratory tract infection (pneumonia), samples tested with Unyvero LRT 55 cartridge and results compared against composite (comparator) which is based on routine clinical microbiology and a second PCR test
  Interventions: Device: LRT55 Testing
- Retrospective Frozen Clinical Specimens: Patients with suspicion of lower respiratory tract infection (pneumonia), samples tested with Unyvero LRT 55 cartridge and results compared against routine clinical microbiology
  Interventions: Device: LRT55 Testing

INTERVENTIONS:
Device: LRT55 Testing — Testing on the Unyvero LRT55

SUMMARY:
The Curetis Unyvero LRT55 Application is intended to detect and to identify genes of 21 microorganisms and 19 genes associated with antibiotic resistance in 4 hours.

In this study, the performance of the Unyvero LRT55 Application shall be tested under clinical conditions and compared to (1) a composite reference method (for non-atypical or cultured microorganisms) or (2) a molecular PCR based reference method for the 3 atypical microorganisms Chlamydophila pneumoniae, Legionella pneumoniae, and Pneumocystis jirovecii, and for resistance genes.

PCR amplifications are followed by bi-directional sequencing, including comparison of the test results Time to result will be compared for the Unyvero LRT55 Application and standard-of care.

DETAILED DESCRIPTION:
This is a non-interventional, controlled, non-randomized multicenter clinical study that compares a new diagnostic device, the Unyvero LRT55 Application (based on molecular diagnostic methods) to either (1) a composite reference method (for non-atypical microorganisms), (2) a composite PCR-based method for 3 atypical microorganisms or (3) a PCR-based reference method for resistance genes.

The study will use leftover lower respiratory tract samples taken from subjects suspected with lower respiratory tract infections: (a) Specimens taken prospectively for standard-of-care (i.e. microbiology testing) from hospitalized subjects. (b) Banked specimens for rare microorganisms.

As the device is under investigation, the test results provided by the Unyvero LRT55 Application will not be made available to the treating physician and therefore will not be used for diagnosis, treatment or other management decisions.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized subjects with suspicion of lower respiratory tract infection
* Age at least 18 years
* Available surplus respiratory aspirate or bronchial lavage sample

Exclusion Criteria:

* Out-patient (ambulatory patient)
* Known infection with HIV, HBV or tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspicion of lower respiratory tract infection in hospitalized subjects.
Sampling Method: Non-Probability Sample
Enrollment: 2124 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Bacher, Study Director — Curetis GmbH
Locations (9):
- United States (9):
  - University of California Los Angeles (UCLA), Los Angeles, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Columbia Universiy Medical Center / New York-Presbyterian Hosp., New York, New York
  - Rochester Medical Center, Rochester, New York
  - Summa Health System, Akron, Ohio
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective Fresh Clinical Specimens | Retrospective Frozen Clinical Specimens
Started | 1653 | 471
Completed | 1653 | 471
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective Fresh Clinical Specimens | Retrospective Frozen Clinical Specimens | Total
Number analyzed (Participants) | 1653 | 471 | 2124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 827 | 186 | 1013
  >=65 years | 826 | 285 | 1111
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 665 | 182 | 847
  Male | 988 | 289 | 1277
Region of Enrollment [Number; unit: participants]
  United States | 1653 | 471 | 2124

OUTCOME MEASURES:

1. Primary Outcome: Clinical Sensitivity and Specificity for Microorganism Detection as Compared to Routine Microbiology and Other Reference Methods Including PCR and Sequencing
Description: Sensitivity for microorganism detection will be determined against the respective reference method consisting of standard procedure and/or a reference method based on PCR and bi-directional sequencing using alternative primers. Sensitivity for non-atypical microorganism detection will thus be determined if at least 1 out of 2 reference methods have identified microorganisms that are covered by the panel of the investigational IVD. Results will further be analyzed against standard of-care alone, as well as against composite comparator. Sensitivity for atypical microorganism detection will be determined against PCR with alternative primers as reference method. Specificity for microorganism detection will be determined in all samples included in the trial. Individual specificities will be calculated for the detection of the respiratory microorganisms analyzed by the investigational IVD compared to the microorganisms reference method.
Time Frame: Up to 12 months
Measure: Mean (95% Confidence Interval); unit: Percentage
Groups:
- Prospective Fresh Clinical Specimens: Patients with suspicion of lower respiratory tract infection (pneumonia), samples tested with Unyvero LRT 55 cartridge and results compared against composite (comparator) which is based on routine clinical microbiology and a second PCR test
  LRT55 Testing: Testing on the Unyvero LRT55
  an overall weighted average sensitivity of 91.4% for detection of panel pathogens an overall weighted average specificity of 99.5% for detection of panel pathogens
  an overall weighted average sensitivity of 89.9 % for detection of resistance markers an overall weighted average specificity of 99.3 % for detection of resistance markers
- Retrospective Frozen Clinical Specimens: Patients with suspicion of lower respiratory tract infection (pneumonia), samples tested with Unyvero LRT 55 cartridge and results compared against routine clinical microbiology
  LRT55 Testing: Testing on the Unyvero LRT55
  an overall weighted average sensitivity of 91.4% for detection of panel pathogens an overall weighted average specificity of 99.5% for detection of panel pathogens
  an overall weighted average sensitivity of 89.9 % for detection of resistance markers an overall weighted average specificity of 99.3 % for detection of resistance markers
Arm/Group | Prospective Fresh Clinical Specimens | Retrospective Frozen Clinical Specimens
Number analyzed (Participants) | 1653 | 471
Percentage
  Sensitivity - Pathogen Detection | 91.4 [91.4 to 91.4] | 91.4 [91.4 to 91.4]
  Specificity- Pathogen Detection | 99.5 [99.5 to 99.5] | 99.5 [99.5 to 99.5]
  Sensitivity - Restistance Marker Detection | 89.9 [89.9 to 89.9] | 89.9 [89.9 to 89.9]
  Specificity - Resistance Marker Detection | 99.3 [99.3 to 99.3] | 99.3 [99.3 to 99.3]

ADVERSE EVENTS:
Description: There were no adverse events monitored or occurring in this study, because this study utilized remnant human biospecimens that had previously been collected for clinical diagnosis not related to the study. All specimens and study testing results were de-identified and had not impact on patient care or treatment.
Arm/Group | Prospective Fresh Clinical Specimens | Retrospective Frozen Clinical Specimens
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No